CLINICAL TRIAL: NCT06391333
Title: Comparison of Supraglottic Airway and Tracheal Intubation on Postoperative Pulmonary Complications Among High-risk Geriatric Patients
Brief Title: Supraglottic Airway vs Tracheal Intubation on PPCs Among High-risk Geriatric Patients
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: RenJi Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: POLMA2
Record Dates: First submitted 2024-04-10; First posted 2024-04-30 (Actual); Last update posted 2024-04-30 (Actual); Status verified 2024-04

CONDITIONS: Pulmonary Complication
Keywords: Supraglottic airway; Tracheal intubation; Postoperative pulmonary complications; Geriatric surgery
MeSH Terms: interventions — Laryngeal Masks

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- laryngeal mask airway (Active Comparator): In this group, patients use a laryngeal mask airway for intraoperative mechanical ventilation.
  Interventions: Device: laryngeal mask airway and endotracheal tube
- endotracheal intubation (Placebo Comparator): In this group, patients use a endotracheal tube for intraoperative mechanical ventilation.
  Interventions: Device: laryngeal mask airway and endotracheal tube

INTERVENTIONS:
Device: laryngeal mask airway and endotracheal tube — The two most commonly used devices for mechanical ventilation.

SUMMARY:
Postoperative pulmonary complications are serious threat to surgical patients, especially to high-risk geriatric patients. There is evidence that laryngeal mask airway is associated with postoperative pulmonary complications in comparison with tracheal intubation. However, conclusion may reverse among frail population such as high-risk geriatric patients. Geriatric patients are often associated with loose mask seal due to physiological changes, which may increase chances of aspiration and pose challenges to intraoperative airway maintenance. It was reported that laryngeal mask airway causes more atelectasis among children, but no report among high-risk elderly. The investigators therefore propose this study to verify the non-inferior effect of laryngeal mask airway compared to tracheal intubation on postoperative pulmonary complications among high-risk geriatric patients undergoing elective non-cardiothoracic surgeries.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged ≥ 70 years scheduled for elective non-cardiothoracic surgery with an ARISCAT score > 44 will be included

Exclusion Criteria:

* Exclusion criteria include emergency surgery; anticipated difficult tracheal intubation; laryngeal pathology that might interfere with supraglottic device insertion; high risk of gastroesophageal reflux; participation in any conflicting trial within the past 3 months; or deemed unsuitable for the trial by investigators.

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 2210 (Estimated)
Dates: Start 2024-05-05 (Estimated); Primary Completion 2026-04-15 (Estimated); Study Completion 2026-06-15 (Estimated)

PRIMARY OUTCOMES:
PPC | 7 days after surgery
  The primary outcome is the incidence of a collapsed composite of postoperative pulmonary complications within 7 postoperative days, diagnosed according to Dr Wang's work published on Anesthesiology, 2022 (PMID: 35226725).

SECONDARY OUTCOMES:
extrapulmonary complications | 7 days after surgery
  extrapulmonary complications according to regular medical reports
severity of PPC | 7 days after surgery
  Clavien Dindo criteria
diagnosis of PPC | 7 days after surgery
  Postoperative pulmonary complications are defined by respiratory infection, respiratory failure, pleural effusion, atelectasis, pneumothorax, bronchospasm, and aspiration pneumonia (Diagnosed according to utcome is the incidence of postoperative pulmonary complications within 7 postoperative days, diagnosed according to Anesthesiology, 2022 (PMID: 35226725).